CLINICAL TRIAL: NCT00508625
Title: A Multicenter, Open Label, Randomized Study of AMG 951 in Subjects With Previously Untreated Stage IIIb/IV Non-Small Cell Lung Cancer (NSCLC) Treated With Chemotherapy With or Without Bevacizumab
Brief Title: A Study of AMG 951 [rhApo2L/TRAIL] in Subjects With Previously Untreated Non-Small Cell Lung Cancer (NSCLC) Treated With Chemotherapy +/- Bevacizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050190
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — TNFSF10 protein, human; Bevacizumab; Carboplatin; Paclitaxel

ARMS (5):
- C (Other): 40 subjects will receive up to 6 cycles of carboplatin (AUC=6.0mg/ml.min) and paclitaxel (200mg/m2) on day 1 of each 21 day cycle plus Bevacizumab (15mg/kg) on day 1 of each 21 day cycle until disease progression, study drug intolerability or withdrawal of consent.
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel
- E (Experimental): 40 subjects will receive up to 6 cycles of carboplatin (AUC=6.0mg/ml.min) and paclitaxel (200mg/m2) on day 1 of each 21 day cycle plus Bevacizumab (15mg/kg) on day 1 and AMG 951 (rhApo2L/TRAIL) (20mg/kg) on days 1-2 per 21 day cycle until disease progression, study drug intolerability or withdrawal of consent.
  Interventions: Drug: AMG 951 (rhApo2L/TRAIL); Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel
- B (Experimental): 40 subjects will receive up to 6 cycles of carboplatin (AUC=6.0mg/ml.min) and paclitaxel (200mg/m2) on day 1 of each 21 day cycle plus AMG 951 (rhApo2L/TRAIL) (8mg/kg) for 5 days per 21 days cycle until disease progression, study drug intolerability or withdrawal of consent.
  Interventions: Drug: AMG 951 (rhApo2L/TRAIL); Drug: Carboplatin; Drug: Paclitaxel
- A (Other): 40 subjects will receive up to 6 cycles of Carboplatin (AUC = 6.0mg/ml.min) and Paclitaxel (200mg/m2) only
  Interventions: Drug: Carboplatin; Drug: Paclitaxel
- D (Experimental): 40 subjects will receive up to 6 cycles of carboplatin (AUC=6.0mg/ml.min) and paclitaxel (200mg/m2) on day 1 of each 21 day cycle plus Bevacizumab (15mg/kg) on day 1 and AMG 951 (rhApo2L/TRAIL) (8mg/kg) on days 1-5 per 21 day cycle until disease progression, study drug intolerability or withdrawal of consent.
  Interventions: Drug: AMG 951 (rhApo2L/TRAIL); Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: AMG 951 (rhApo2L/TRAIL) — AMG 951 is recombinant human Apo2Ligand/Tumor necrosis factor related apoptosis inducing ligand (rhApo2L/TRAIL) that triggers apoptosis through activation of death receptor 4 (DR4) and death receptor 5 (DR5).
  Other Names: Dulanermin
  Arms: B; D; E
Drug: Bevacizumab — Bevacizumab is a recombinant humanized version of a murine antibody to vascular endothelial growth factor (VEGF).
  Other Names: Avastin
  Arms: C; D; E
Drug: Carboplatin — Standard platinum based chemotherapy
Drug: Paclitaxel — Standard taxane chemotherapy

SUMMARY:
This is a phase 2 multicenter, open label, randomized study of AMG 951 (rhApo2L/TRAIL) in subjects with previously untreated stage IIIb/IV NSCLC treated with chemotherapy with or without bevacizumab.

Subjects will be assigned to a set of treatment groups depending on their eligibility to receive bevacizumab. Subjects with squamous NSCLC and/or CNS metastases will not be eligible to receive bevacizumab and will be assigned to either cohort A or B (provided all other eligibility criteria are met). Subjects who are eligible to receive bevacizumab will be assigned to cohort C, D or E. Cohorts are defined as follows:

Subjects with squamous NSCLC or CNS mets:

Cohort A: Chemotherapy alone Cohort B: Chemotherapy plus 8 mg/kg AMG 951 for 5 days

Subjects without squamous NSCLC and without CNS mets:

Cohort C: Chemotherapy and bevacizumab Cohort D: Chemotherapy, bevacizumab plus 8 mg/kg AMG 951 for 5 days Cohort E: Chemotherapy, bevacizumab plus up to 20 mg/kg AMG 951 for 2 days Approximately forty subjects will be recruited to each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Non-Small Cell Lung Cancer (NSCLC). Mixed tumors will be categorized by the predominant cell type unless small cell elements are present in which case the patient is ineligible. Cytologic or histologic elements can be established on metastatic tumor aspirates or biopsy.
* Subjects must have advanced NSCLC defined as stage IIIb with malignant pleural effusion or Stage IV or recurrent disease. Subjects with unmeasurable but evaluable disease can be included in the phase 1b study, but disease must be measurable to be included in the phase 2 study
* Planning to receive up to 6 cycles of chemotherapy
* ECOG performance status of 0 or 1
* Life expectancy greater than 3 months
* ≥18 years old
* Subjects must sign and date a written Independent Ethics Committee (IEC)-approved Informed Consent Form
* INR ≤ 1.2 and PTT ≤ ULN within 1 week prior to enrollment

Exclusion Criteria:

Disease Related

* Prior malignancy other than NSCLC (except in situ basal cell carcinoma or in situ cervical cancer), unless have been treated with curative intent with no evidence of disease for > 3 years
* Untreated or unstable central nervous system (CNS) metastases. Subjects with treated and stably controlled CNS metastases are eligible for cohorts A and B of the phase 2 part of the study if definitive therapy has been administered (surgery and/or radiation therapy), there is no planned treatment for brain metastases, and the subject is clinically stable and is off corticosteroids or on a stable dose of corticosteroids for at least 2 weeks prior to enrollment
* Myocardial infarction, or unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure [New York Heart Association > class II]) within 1 year of enrollment
* Uncontrolled hypertension defined as: systolic blood pressure > 150 mm Hg OR diastolic blood pressure > 100 mm Hg (antihypertensive therapy to achieve these parameters is allowable)
* History of arterial thrombosis, pulmonary embolus, deep vein thrombosis or hemorrhagic disorders within 1 year of enrollment
* Recent major surgical procedure within 28 days of enrollment
* Subjects must not have serious non-healing wound ulcer, or bone fracture within 21 days prior to enrollment
* Persistent history of gross hemoptysis (defined as bright red blood of a ½ teaspoon or more) related to subject's NSCLC
* Known (documented in medical notes) HIV infection
* Active infection on day of enrollment
* Known to be hepatitis C positive OR hepatitis B surface antigen positive
* Subjects with Gilbert's syndrome

Laboratory

* Absolute neutrophil count (ANC) < 1.5 x 10*9 /L (without granulocyte-colony stimulating factor support within 2 weeks of enrollment)
* Platelet count < 100 x 10*9 /L (without transfusion within 2 weeks of enrollment)
* Hemoglobin < 9 g/dL (subjects may be transfused or receive erythropoietic treatment to meet criterion)
* Urine protein quantitative value of > 1+ on dipstick or > 30 mg/dL in urinalysis. If quantitative protein is < 500 mg in 24-hour urine collection then subject can be included
* Significant liver dysfunction as defined by aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x upper limits of normal (ULN)
* Alkaline phosphatase > 2.5 x ULN, or alkaline phosphatase > 5 x ULN in the presence of bone or liver metastasis
* Total bilirubin > 1.5 x ULN
* Calculated creatinine clearance < 50 mL/min.
* Hypercalcemia (serum calcium > 12.0 mg/dL or symptomatic)

Medications

* Prior chemotherapy (except for adjuvant chemotherapy, provided the last dose of adjuvant therapy was received at least one year prior to enrollment), hormonal therapy, radiotherapy (except palliative radiotherapy for bone metastases or radiation therapy for CNS metastases) or immunotherapy for treatment of advanced NSCLC
* Prior drug treatment or therapy with investigational agents for NSCLC
* Therapeutic anticoagulation treatment. Prophylactic anticoagulation of venous access devices (eg, with low-dose warfarin [1-2mg/day] or low-dose heparin) is allowed providing INR ≤ 1.2 and PTT is ≤ ULN within 1 week prior to enrollment
* Chronic daily treatment with aspirin (> 325 mg/day) or non-steroidal anti-inflammatory agents known to inhibit platelet function. Treatment with dipyridamole, ticlopidine, clopidogrel and/or cilostazol is also not allowed.

General Exclusions

* Participation in clinical trials or undergoing other investigational procedures within 30 days before study enrollment
* Subject is evidently pregnant (e.g. positive HCG test) or is breast feeding
* Woman or man with partner of childbearing potential not consenting to use adequate contraceptive precautions i.e. double barrier contraceptive methods (eg diaphragm plus condom), or abstinence during the course of the study and for 6 months after the last study drug administration for women, and 1 month for men.
* Subject has known sensitivity to any of the products to be administered during the study.
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or comply with study procedures.
* Any condition which in the investigator's opinion makes the subject unsuitable for study participation
* Subjects enrolled and dosed in phase 1b will be excluded from phase 2

Exclusion criteria for phase 1b and bevacizumab treatment (cohorts C, D and E) in phase 2

* Subjects with central nervous system tumor involvement
* Subjects with squamous NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate (CR and PR) by modified RECIST | Until disease progression, drug intolerability or withdrawal of consent

SECONDARY OUTCOMES:
Progression free survival | Until disease progression, drug intolerability or withdrawal of consent
Time to response | Until disease progression, drug intolerability or withdrawal of consent
Duration of response | Until disease progression, drug intolerability or withdrawal of consent
Time to progression | Until disease progression, drug intolerability or withdrawal of consent
Overall response rate (complete, partial or stable response) | Until disease progression, drug intolerability or withdrawal of consent
Overall Survival | Until disease progression, drug intolerability or withdrawal of consent

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Besse B, Planchard D, Veillard AS, Taillade L, Khayat D, Ducourtieux M, Pignon JP, Lumbroso J, Lafontaine C, Mathiot C, Soria JC. Phase 2 study of frontline bortezomib in patients with advanced non-small cell lung cancer. Lung Cancer. 2012 Apr;76(1):78-83. doi: 10.1016/j.lungcan.2011.09.006. Epub 2011 Dec 18. PMID 22186627
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com